CLINICAL TRIAL: NCT02907047
Title: Tourniquet vs. no Tourniquet During Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Model: Parallel
Other Study IDs: 16Austin01
Record Dates: First submitted 2016-09-15; First posted 2016-09-20 (Estimated); Last update posted 2019-07-01 (Actual); Status verified 2019-06

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

ARMS (2):
- Tourniquet (Active Comparator): These subjects will have their tourniquet inflated during key portions of the total knee arthroplasty procedure
  Interventions: Other: tourniquet inflated
- No tourniquet (Other): These subjects will not have their tourniquet inflated during key portions of the total knee arthroplasty procedure
  Interventions: Other: tourniquet not inflated

INTERVENTIONS:
Other: tourniquet inflated
  Arms: Tourniquet
Other: tourniquet not inflated
  Arms: No tourniquet

SUMMARY:
The purpose of this study is to correlate functional outcomes and perioperative complications with tourniquet use during total knee arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

1. All unilateral primary knee arthroplasties performed by investigators participating in this study will be eligible for inclusion
2. Diagnosis of osteoarthritis

Exclusion Criteria:

1. Revision surgery
2. Bilateral knee surgery
3. Age <18 or >80
4. BMI >40
5. Baseline lower extremity strength less than 5/5
6. Vascular calcifications
7. History of chronic narcotic use, defined as more than 5mg of oxycodone q4 hours
8. Functionally limiting spine disease
9. Other functionally limiting lower extremity disorder (i.e. symptomatic ipsilateral hip disease)
10. Patients who cannot perform the baseline functional tests
11. Allergy/contraindication to protocol medications
12. Post-traumatic arthritis
13. Inflammatory arthritis
14. Pregnancy
15. Prisoners
16. Patients receiving care as part of a worker's compensable injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2016-06-01 (Actual); Primary Completion 2017-04-01 (Actual); Study Completion 2017-10-01 (Actual)

PRIMARY OUTCOMES:
timed up and go (TUG) score | 4 weeks following surgery
Stair Climb test | in hospital (usually less than 2 days), 4 weeks post-op, 6 months post-op
  time, in seconds, to climb one flight of nine stairs
Visual Analog Scale: Pain | in hospital (usually less than 2 days), 4 weeks post-op, 6 months post-op

SECONDARY OUTCOMES:
blood loss | intra-operative
  calculated blood loss determine by hemoglobin dilution
surgical field visualization | intra-operative
  subjective rating provided by the surgeon
range of motion | in hospital (usually less than 2 days), 4 weeks post-op, 6 months post-op
  measured, in degrees, using a goniometer

CONTACTS AND LOCATIONS:
Locations (1):
- Rothman Institute, Philadelphia, Pennsylvania, United States